CLINICAL TRIAL: NCT00000296
Title: Role of Metabolites in Nicotine Dependence (4)
Brief Title: Role of Metabolites in Nicotine Dependence (4) - 13
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-13; P50-09259-13
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1999-02

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Drug: Cotinine fumarate

SUMMARY:
The purpose of this study is to determine the effects of cotinine with or without a transdermal nicotine replacement on tobacco withdrawal symptoms.

DETAILED DESCRIPTION:
Previous studies have shown that cotinine, a metabolite of nicotine, antagonizes some of the effects of nicotine. One study showed that nicotine eliminates some of the beneficial effects of the nicotine patch in reducing withdrawal symptoms. The purpose of this study was to replicate and extend these findings and examine the effects of various doses of cotinine base compared placebo on withdrawal symptom as well as drug preference among abstinent smokers while using the nicotine patch. We hypothesized that cotinine will reduce the beneficial effects of the nicotine patch in reducing withdrawal symptoms and that placebo will be preferred over cotinine during the forced drug choice period.

ELIGIBILITY:
Inclusion Criteria:

Male/Female subjects, aged 21-45 years inclusive, with a smoking history of at least 20 cigarettes daily (greater than or equal to 50) for at lease 1 year. Subject is in good health as verified by medical history, screening examination, and screening laboratory tests as outlined above. Subject has provided written informed consent to participate in the study and is motivated to stop smoking. Subject has experienced at least 4 withdrawal symptoms upon abstinence.

Exclusion Criteria:

History of myocardial infarction, angina pectoris, sustained or episodic cardiac arrhythmias, symptomatic peripheral vascular disease, current peptic ulcer disease or any other medical condition which the physician investigator deems inappropriate for subject participation. Insulin-dependent diabetes. Pregnant or lactating, or not using adequate birth control methods. Requirement of any form of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric history (less than 1yr). Chronic use of systemic steroids or antihistamines. Abuse of alcohol or any other recreation aor prescription drug (more tha 3 drinks per day or 21 drinks per week). Use of any other nicotine products, including smokeless tobacco, cigars and nicotine replacement products. Inability to fulfill all scheduled visits and examination procedures throughout the study period. History of schizophrenia or manic depressive disorder. Recent history of other psychiatric illness;less than 1 year since last episode of major depressive episode.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1997-11; Study Completion 2001-12

PRIMARY OUTCOMES:
Subjective effects
Physiological effects
Behavioral

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Presented at Society for Research on Nicotine: Tobacco. None